CLINICAL TRIAL: NCT05985785
Title: Bone Marrow Aspirate Concentrate vs Corticosteroid Injection for Symptomatic Osteoarthritis (OA) of the Knee: A Randomized Controlled Trial
Brief Title: Bone Marrow Aspirate Concentrate (BMAC) vs Corticosteroid Injection
Acronym: BMAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21052504
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Treatment arms include BMAC injections (ARM1) and corticosteroid injections (ARM 2). Patients in the corticosteroid injection group (ARM 2) will receive a sham incision. Follow-up will be up to six months (12-months if crossover (ARM 3)).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autologous (from subject to self) bone marrow aspirate concentrate (BMAC) injections (Experimental): Autologous bone marrow aspirate concentrate (BMAC) will be removed from the subject knee body with a needle, processed and concentrated by an FDA-approved centrifuge (separator) system. The concentrated cells will be injected into the subject knee. "Autologous" means that the subject is receiving back their own cells that were collected.
  Interventions: Other: Autologous bone marrow aspirate concentrate (BMAC)
- Corticosteroid injection (Active Comparator): Corticosteroid injection group (ARM 2) will receive a sham incision.
  Interventions: Drug: Corticosteroid injections
- Crossover Group (Other): Any patient in the corticosteroid injection group that shows no improvement in pain after 24 weeks (12 month follow-up if crossover), per physician discretion, will be allowed crossover to the BMAC injection group (ARM 3).
  Interventions: Other: Crossover Autologous bone marrow aspirate concentrate (BMAC)

INTERVENTIONS:
Other: Autologous bone marrow aspirate concentrate (BMAC) — Bone marrow aspirate concentrate BMAC is a biologically substance harvested from a patient for autologous use. Bone marrow aspirate concentrate (BMAC) has been determined by the FDA to be a minimally manipulated biologic prepared for autologous use and does not require premarket FDA approval for clinical use.
  Arms: Autologous (from subject to self) bone marrow aspirate concentrate (BMAC) injections
Drug: Corticosteroid injections — Current standard of treatment for OA of the knee is corticosteroid injection.
  Arms: Corticosteroid injection
Other: Crossover Autologous bone marrow aspirate concentrate (BMAC) — Subjects who participate in this study and who are randomized to receive the BMAC may experience decreased pain and increased functionality after the injection compared to those that receive a corticosteroid injection. As such, participants who continue to have pain after a corticosteroid injection will be allowed to crossover to a BMAC injection at 24 weeks or 6 months post-surgery.(ARM 3)
  Arms: Crossover Group

SUMMARY:
Prospective single-masked (study participant will be masked), randomized controlled trial to examine the influence of BMAC on patient-reported outcomes (PROs) in patients with primary knee osteoarthritis.

DETAILED DESCRIPTION:
The purpose of this study is to examine the influence of BMAC on patient-reported outcomes (PROs) in patients with primary knee osteoarthritis and compare that to patients receiving corticosteroid injections with six-month follow-up.

All patients who sign the consent form will be enrolled in the study and randomized to one of the two treatment arms. This study will aim to recruit and enroll a total of 100 patients (50 per group). Treatment arms include BMAC injections (ARM1) and corticosteroid injections (ARM 2). Patients in the corticosteroid injection group (ARM 2) will receive a sham incision. Follow-up will be up to six months (12-months if crossover (ARM 3)).

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-70
* Long standing knee pain from osteoarthritis (KL grade 2-3) despite conventional treatments such as activity modification, weight loss, physical therapy, analgesics, nonsteroidal anti-inflammatory drugs, or injection therapy for at least 6 weeks
* 7-day average pain score of at least 4 on VAS scale

Exclusion Criteria:

* Systemic diseases (Diabetes, malignancies, infections, etc.)
* Post-traumatic arthritis
* Patient had intra-articular injection on affected knee in last three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) for pain | Enrollment up to 6 months postoperatively (12 months if crossover from ARM 3 to ARM 1)
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.
Intermittent and Constant Osteoarthritis Pain (ICOAP) | Enrollment up to 6 months postoperatively (12 months if crossover from ARM 3 to ARM 1)
  13 items survey that assess two forms of pain reported by people with osteoarthritis: intermittent and constant pain.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Enrollment up to 6 months postoperatively (12 months if crossover from ARM 3 to ARM 1)
  The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Chahla, MD, Principal Investigator — Rush University Medical Center Associate Professor and Surgeon
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States